CLINICAL TRIAL: NCT07311733
Title: Milky Way Sensor: Device Validation for Infiltrated Tissues
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVW-CLR-CS38-400
Record Dates: First submitted 2025-12-29; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Infiltration of Peripheral IV Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Infiltrated Tissue (Experimental): The ivWatch Milky Way sensors monitored an IV site during the infiltration of 10 mL of isotonic saline solution. IV sites were placed in the forearm and the dorsal aspect of the hand. The rate of the infiltration ranged between 5 mL/hr to 150 mL/hr.
  Interventions: Device: ivWatch Model 400 with Milky Way Sensor

INTERVENTIONS:
Device: ivWatch Model 400 with Milky Way Sensor — The ivWatch Model 400 with Milky Way Sensor monitored the site during the course of the infiltration and issued red and/or yellow notifications if an infiltration was detected.

SUMMARY:
A single arm trial consisting of 28 adult volunteers to assess the safety and efficacy of ivWatch sensors when observing infiltrated tissues at common sites for peripheral IV therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Healthy, verified by an eligible designation on the Health History Form

Exclusion Criteria:

* Abnormal bleeding / hemophilia
* Absence of sensation in one or both arms
* Allergy to common medical materials
* Blood clotting disorder
* Currently enrolled in another clinical trial
* Current hepatitis infection or any history of hepatitis B or C
* Currently pregnant
* Daily regimen of blood thinning medication (e.g., aspirin, ibuprofen, naproxen, Coumadin®/warfarin, Eliquis®/apixaban).
* Fever at the time of study visit (≥100.4°F)
* Frequent dizziness or fainting spells, especially with needles
* History of chronic, severe anemia
* History of stroke
* HIV / Aids
* Immune deficiency disorder
* Lymphedema
* Major surgery or scar tissue which would complicate PIV access
* Needle phobia
* Radiation / chemotherapy in the last year
* Received IV therapy in 14 days prior to study visit
* Severe dehydration on day of study visit
* Sick or had an infection in 14 days prior to study visit
* Tattoo(s) that severely limits vein visualization at a sensor monitoring location
* Unstable or uncontrolled cardiopulmonary disorder
* Uncontrolled seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Red Notification Sensitivity to Infiltrated Tissues | After each participant has been infiltrated, an expected average of 1 hour.
  The ratio of the number of infiltrated IV sites where the ivWatch Model 400 device issued a red notification to the total number of infiltrated IV sites in the study. All infiltrations were limited to 10 mL of isotonic saline solution.

SECONDARY OUTCOMES:
Yellow Notification Sensitivity to Infiltrated Tissues | After each participant has been infiltrated, an expected average of 1 hour.
  The ratio of the number of infiltrated IV sites where the ivWatch Model 400 device issued a yellow notification to the total number of infiltrated IV sites in the study. All infiltrations were limited to 10 mL of isotonic saline solution.
Significant Skin Irritation or Disruption to Skin Integrity | After each participant has been infiltrated, an expected average of 1 hour.
  The number of IV sites that indicated significant skin irritation or disruption to skin integrity assessed at the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- ivWatch, Newport News, Virginia, United States